CLINICAL TRIAL: NCT02240407
Title: Evaluation of Re-administration of Recombinant Adeno-Associated Virus Acid Alpha-Glucosidase (rAAV9-DES-hGAA) in Patients With Late-Onset Pompe Disease (LOPD)
Brief Title: Re-administration of Intramuscular AAV9 in Patients With Late-Onset Pompe Disease
Acronym: AAV9-GAA_IM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Lacerta Therapeutics (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB201400137; 20182574 (Other: WIRB)
Record Dates: First submitted 2014-09-11; First posted 2014-09-15 (Estimated); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Pompe Disease
Keywords: Pompe Disease; Gene Therapy; Repeated dosing; Immune modulation
MeSH Terms: conditions — Glycogen Storage Disease Type II | interventions — Sirolimus; Sodium Chloride; Excipients; Rituximab; Diphenhydramine; Acetaminophen; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- rAAV9-DES-hGAA vector (Experimental): Each subject will receive Rituxan and Rapamycin prior to the initial exposure to the study agent in one leg and the subsequent exposure of the same vector to the contralateral leg after four months. Diphenhydramine and acetaminophen will be provided before each Rituxan dose. Immune Globulin will be administered to each subject every other month after first exposure to Rituxan and as clinical necessary. Lidocaine will be administered through percutaneous infiltration before injection of the study agent. Side of administration will be randomized at first Recombinant Adeno-Associated Virus Acid Alpha-Glucosidase injection.
  Interventions: Genetic: Recombinant Adeno-Associated Virus Acid Alpha-Glucosidase; Drug: Rapamycin; Drug: Rituxan; Drug: Diphenhydramine; Drug: Acetaminophen; Drug: Lidocaine; Drug: LMX 4 Topical Cream
- Excipient (Sham Comparator): Each subject will receive Rituxan and Rapamycin prior to the initial exposure to the study agent in one leg and the subsequent exposure of the same vector to the contralateral leg after four months. Diphenhydramine and acetaminophen will be provided before each Rituxan dose. Immune Globulin will be administered to each subject every other month after first exposure to Rituxan and as clinical necessary. Lidocaine will be administered through percutaneous infiltration before injection of the study agent. Side of administration will be randomized at first saline injection.
  Interventions: Drug: Rapamycin; Other: saline; Drug: Rituxan; Drug: Diphenhydramine; Drug: Acetaminophen; Drug: Lidocaine; Drug: LMX 4 Topical Cream

INTERVENTIONS:
Genetic: Recombinant Adeno-Associated Virus Acid Alpha-Glucosidase — The dose selected for this study is a fixed dose of 4.6 x 10^13 vg per TA muscle (range of 7.64 x 10^11 vg/gm to 4.6 x 10^11 vg/gm based on TA weight).
  Other Names: rAAV9-DES-hGAA
  Arms: rAAV9-DES-hGAA vector
Drug: Rapamycin — Patients will receive Rapamycin (dose 0.6-2 mg/m^2/day, adjusted to maintain a trough serum sirolimus level of 2-4 ng/mL.) every day starting from 7 days before first injection of AAV9 until four months after second injection.
  Other Names: Sirolimus
Other: saline — Same volume as rAAV9-DES-hGAA injection will be used.
  Other Names: Excipient
  Arms: Excipient
Drug: Rituxan — Patients will receive Rituxan (dose: 750 mg/m^2 twice) 21 and 7 day prior first AAV9 injection, with a Rituxan dose 375 mg/m^2 on the day of the injection. Rituxan will be repeated 7 days prior to the 2nd injection of the vector. The maintenance dose of Rituxan will be 375 mg/m^2.
  Other Names: Rituximab
Drug: Diphenhydramine — 25-50mg will be provided before each Rituximab dose.
  Other Names: Benadryl
Drug: Acetaminophen — We will provide 650 mg of tylenol before each dose of Rituximab.
  Other Names: Tylenol
Drug: Lidocaine — Lidocaine will be used based on standard of care: Percutaneous infiltration, concentration 0.5-1%, 1-10 mL, 5-300mg total dose.
  Other Names: Xylocaine
Drug: LMX 4 Topical Cream — Topical anesthesia cream will be used prior to gene therapy/saline injection.
  Other Names: Lidocaine 4%

SUMMARY:
A recombinant AAV vector has been generated to carry the codon-optimized acid alpha-glucosidase (coGAA) gene expressed from a human desmin enhancer/promoter (DES). The proposed clinical trial is a within-participant, double-blind, randomized, phase I controlled study evaluating the toxicology, biodistribution and potential activity of re-administration of rAAV9-DES-hGAA injected intramuscularly into the TA. Nine participants (18 to 50-years old) who reside within the United States with Late-Onset Pompe Disease (LOPD) will be included. The goal of the immune modulation strategy is to ablate B-cells (Rituximab and Sirolimus) prior to the initial exposure to the study agent in one leg and the subsequent exposure of the same vector to the contralateral leg after four months. At each study agent dosing, the contralateral leg will receive excipient. Patients will act as their own controls. Repeated measures, at baseline and during the following 3 months after each injection, will assess the safety, biochemical and functional impact of the vector.

DETAILED DESCRIPTION:
Enrolling in this study will entail participating in 18 months of study-related visits. Patients will be asked to come to the Clinical and Translational Research Building at the University of Florida for a series of onsite study visits.

All the visits will be performed as outpatient procedures at the Clinical Research Center (CRC) and at other facilities at the University of Florida. Overnight observation will not be needed, however, patients will be asked to stay overnight in a hotel near the University of Florida. During the first 4 months after each injection, patients will be asked to perform outpatient laboratory work at a laboratory facility convenient for them.

In addition, during this study patients will be asked to take medications that will modulate the ability of their immune system to react against foreign agents including the gene transfer agent. The purpose of these medications is to improve the activity of the GAA within the body. Patients will receive a Rituximab injection 21 days prior to the first injection of the study agent and 7 days before each injection of the study agent and the day of the first injection. Rituximab will be delivered by infusion that may last 2-6 hours. Patients will need to take another medication (Sirolimus) every day starting 7 days before the first injection of the study agent until four months after the second injection of the study agent.

The following discusses what will occur at each visit:

Baseline Baseline Evaluation and first Rituximab infusion - Day -22/-21/-20

* Medical history: Patients will be asked to complete a questionnaire about his/her medical history.
* Physical exam: The study doctor will perform a general physical exam to evaluate patients physical health.
* Blood and urine tests: These tests will be used for evaluating the safety of the gene transfer agent.
* Electrocardiogram (ECG): This test will measure the electrical activity of patient's heart to see if it is working properly.
* Quantitative Muscle Testing (QMT): This test finds out how strong the patient's leg muscles are.
* 10 Meter Walk Test: Patients will be instructed to walk a set distance (10 meters); time will be measured while patient walks the set distance and the distance covered will be divided by the time it took to walk that distance.
* Gait analysis: Gait will be tested with Gait Mat II, which will record the spatial and temporal parameters of his/her walk such as cadence, speed and distance between your feet.
* Magnetic Resonance Imaging (MRI) and Spectroscopy (MRS): MRI and MRS testing will be done inside a large magnet that lets the study doctors measure the size and health of the patient's muscles. These tests are done at the same time. MRI and MRS testing will require the patient to stay very still for up to an hour.
* Magnetic stimulation of the common fibular nerve: The common fibular nerve, which is the nerve that controls the injected muscle, will be stimulated with a magnetic field to test the impact of the gene transfer agent to the nervous system.
* The patient will receive the first Rituximab infusion. It might last between 2 and 6 hours.

Rituximab infusion - Day -6

* The patient will receive the 2nd Rituximab infusion 7 days before the gene transfer agent. It might last between 2 and 6 hours.
* Patient will begin Rapamycin.

  1st Injection - Day 0/1
* The patient will receive the 3rd Rituximab infusion the day before the gene transfer agent. It might last between 2 and 6 hours.
* Patient will receive the gene transfer agent in 1 injection (a total of about 1 teaspoon) into the tibialis anterior (TA) muscle of one leg. The other leg will receive a pharmacologically inactive solution. An ultrasound will be used to detect the proper location of injection. A photograph of the injection at the injection site may be taken. If the patient agrees to this, he/she will be asked to sign a consent form for this procedure.

On day 1, blood tests will be done.

Outpatient lab work - Day 3/7/15/30/60

* Blood and urine tests

Onsite visit - Day 89/90

* Medical history
* Physical Exam
* Blood and urine tests
* Quantitative Muscle Testing (QMT)
* 10 Meter Walk Test
* Gait analysis
* Magnetic Resonance Imaging (MRI) and Spectroscopy (MRS)
* Muscle Biopsy: Tissue samples obtained will be used for evaluation of muscle glycogen and GAA activity in the injected muscle.
* Magnetic stimulation of the common fibular nerve

Rituximab infusion - Day 114

* The patient will receive the 4th Rituximab infusion, it might last between 2-6 hours.

  2nd Injection - Day 121/122
* The patient will receive the second gene transfer agent injection in the leg that previously received the inactive solution. The leg that previously received the study agent will receive the inactive solution. The injection procedure and the amount of study agent injected will be the same as the first injection.

On day 122, blood tests will be done.

Outpatient lab work - Day 124/128/135/150/180

* Blood and urine tests

Onsite visit - Day 209/210

* Medical History
* Physical Exam
* Blood and urine tests
* Quantitative Muscle Testing (QMT)
* 10 Meter Walk Test
* Gait analysis
* Magnetic Resonance Imaging (MRI) and Spectroscopy (MRS)
* Muscle Biopsy
* Magnetic stimulation of the common fibular nerve

Onsite visit - Day 365

* Medical history
* Physical exam
* Quantitative Muscle Testing (QMT)
* 10 Meter Walk Test
* Blood and urine tests

Onsite visit - Day 520

* Medical history
* Physical exam
* Quantitative Muscle Testing (QMT)
* 10 Meter Walk Test
* Blood and urine tests

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 18 to 50-years old
* Have a diagnosis of Pompe disease, as defined by protein assay AND/OR DNA sequence of the acid alpha-glucosidase gene, AND clinical symptoms of the disease
* Have residual ability to complete the 10 meter walk test
* Willing to discontinue aspirin, aspirin-containing products and other drugs that may alter platelet function, 7 days prior to dosing, resuming 24 hours after the dose has been administered
* Consistently taking enzyme replacement therapy (ERT) or remain off ERT from baseline until Day 520
* United States residents only.

Exclusion Criteria:

* Be pregnant or nursing, and if the subject is of child bearing potential they should use contraception until the end of the study
* Have required oral or systemic corticosteroids within the last 15 days prior to baseline screening
* Have a platelet count less than 75,000/mm^3
* Have an INR greater than 1.3
* Have seronegative to AAV9 capsid protein (neutralizing Ab titers <1:5 and total binding Ab titer <50 U/ml)
* Have transaminases and alkaline phosphatase more than ten times the upper limit of normal at screening or Day-1
* Have bilirubin and gamma-glutamyl transpeptidase greater than 2 times the upper limit of normal at screening or Day -1
* Have any chronic liver disease (aside from hepatic dysfunction related to Pompe disease) such as hepatitis B and C and cirrhosis
* Be currently, or within the past 30 days, participating in any other research protocol involving investigational agents or therapies
* Have history of platelet dysfunction, evidence of abnormal platelet function at screening, or history of recent use of drugs that may alter platelet function, which the subject is unable/unwilling to discontinue for study agent administration
* Have received gene transfer agents within the past 6 months
* Have any medical condition or circumstance for which an MRI evaluation is contraindicated
* Have any other concurrent condition that, in the opinion of the investigator, would make the subject unsuitable for the study
* Inconsistent with use of ERT.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2017-10-17 (Actual); Primary Completion 2021-08-26 (Actual); Study Completion 2021-08-26 (Actual)

PRIMARY OUTCOMES:
Safety of rAAV9-DES-hGAA vector in LOPD by blood and urine test. | 520 days
  Safety will be tested by clinical pathology tests, blood assay for vector genomes, antibodies against GAA and T-cell ELISPOT against GAA and AAV.

SECONDARY OUTCOMES:
Neurophysiological tests will be performed for neuro function of rAAV9-DES-hGAA vector. | 520 days
  Neurophysiological tests: Surface testing of the common fibular nerve and neuromuscular junction transmission.
Muscle biopsy will be performed for muscular function of rAAV9-DES-hGAA vector. | 520 days
  Muscle biopsy for biochemistry and immunochemistry tests.
Clinical tests will be performed for function of rAAV9-DES-hGAA vector. | 520 days
  Clinical tests: 10 meter walk test and muscle strength test.
Magnetic Resonance Imaging will be performed for visualization of muscle with rAAV9-DES-hGAA vector. | 520 days
  MRI will provide a non-invasive means of evaluating maximum cross-sectional area (CSAmax) - an index of muscle mass - and the MR proton traverse relaxation time (T2) - an index of muscle damage and edema.
Spectroscopy will be performed for function of rAAV9-DES-hGAA vector. | 520 days
  MRS will provide a non-invasive means of evaluating glycogen concentration in muscle.

CONTACTS AND LOCATIONS:
Overall Officials: Manuela Corti, P.T., PhD., Principal Investigator — University of Florida
Locations (1):
- Clinical and Translational Research Building (CTRB), University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Corti M, Smith BK, Falk DJ, Lawson LA, Fuller DD, Subramony SH, Byrne BJ, Christou EA. Altered activation of the tibialis anterior in individuals with Pompe disease: Implications for motor unit dysfunction. Muscle Nerve. 2015 Jun;51(6):877-83. doi: 10.1002/mus.24444. Epub 2015 Apr 24. PMID 25186912
- [Background] McKusick V. 232300 Glycogen Storage Disease II. OMIM. 1996.
- [Background] Moufarrej NA, Bertorini TE. Respiratory insufficiency in adult-type acid maltase deficiency. South Med J. 1993 May;86(5):560-7. doi: 10.1097/00007611-199305000-00015. PMID 8488406
- [Background] Wokke JH, Escolar DM, Pestronk A, Jaffe KM, Carter GT, van den Berg LH, Florence JM, Mayhew J, Skrinar A, Corzo D, Laforet P. Clinical features of late-onset Pompe disease: a prospective cohort study. Muscle Nerve. 2008 Oct;38(4):1236-45. doi: 10.1002/mus.21025. PMID 18816591
- [Background] Byrne BJ, Falk DJ, Pacak CA, Nayak S, Herzog RW, Elder ME, Collins SW, Conlon TJ, Clement N, Cleaver BD, Cloutier DA, Porvasnik SL, Islam S, Elmallah MK, Martin A, Smith BK, Fuller DD, Lawson LA, Mah CS. Pompe disease gene therapy. Hum Mol Genet. 2011 Apr 15;20(R1):R61-8. doi: 10.1093/hmg/ddr174. Epub 2011 Apr 25. PMID 21518733
- [Background] Byrne BJ, Kishnani PS, Case LE, Merlini L, Muller-Felber W, Prasad S, van der Ploeg A. Pompe disease: design, methodology, and early findings from the Pompe Registry. Mol Genet Metab. 2011 May;103(1):1-11. doi: 10.1016/j.ymgme.2011.02.004. Epub 2011 Feb 11. PMID 21439876
- [Background] Lee KZ, Qiu K, Sandhu MS, Elmallah MK, Falk DJ, Lane MA, Reier PJ, Byrne BJ, Fuller DD. Hypoglossal neuropathology and respiratory activity in pompe mice. Front Physiol. 2011 Jun 30;2:31. doi: 10.3389/fphys.2011.00031. eCollection 2011. PMID 21747768
- [Background] Benowitz LI, Routtenberg A. GAP-43: an intrinsic determinant of neuronal development and plasticity. Trends Neurosci. 1997 Feb;20(2):84-91. doi: 10.1016/s0166-2236(96)10072-2. PMID 9023877
- [Background] Kanazir S, Ruzdijic S, Vukosavic S, Ivkovic S, Milosevic A, Zecevic N, Rakic L. GAP-43 mRNA expression in early development of human nervous system. Brain Res Mol Brain Res. 1996 May;38(1):145-55. doi: 10.1016/0169-328x(96)00008-3. PMID 8737678
- [Background] Vilchez D, Ros S, Cifuentes D, Pujadas L, Valles J, Garcia-Fojeda B, Criado-Garcia O, Fernandez-Sanchez E, Medrano-Fernandez I, Dominguez J, Garcia-Rocha M, Soriano E, Rodriguez de Cordoba S, Guinovart JJ. Mechanism suppressing glycogen synthesis in neurons and its demise in progressive myoclonus epilepsy. Nat Neurosci. 2007 Nov;10(11):1407-13. doi: 10.1038/nn1998. Epub 2007 Oct 21. PMID 17952067
- [Background] DeRuisseau LR, Fuller DD, Qiu K, DeRuisseau KC, Donnelly WH Jr, Mah C, Reier PJ, Byrne BJ. Neural deficits contribute to respiratory insufficiency in Pompe disease. Proc Natl Acad Sci U S A. 2009 Jun 9;106(23):9419-24. doi: 10.1073/pnas.0902534106. Epub 2009 May 27. PMID 19474295
- [Background] Foust KD, Nurre E, Montgomery CL, Hernandez A, Chan CM, Kaspar BK. Intravascular AAV9 preferentially targets neonatal neurons and adult astrocytes. Nat Biotechnol. 2009 Jan;27(1):59-65. doi: 10.1038/nbt.1515. Epub 2008 Dec 21. PMID 19098898
- [Background] Weinstein DA, Correia CE, Conlon T, Specht A, Verstegen J, Onclin-Verstegen K, Campbell-Thompson M, Dhaliwal G, Mirian L, Cossette H, Falk DJ, Germain S, Clement N, Porvasnik S, Fiske L, Struck M, Ramirez HE, Jordan J, Andrutis K, Chou JY, Byrne BJ, Mah CS. Adeno-associated virus-mediated correction of a canine model of glycogen storage disease type Ia. Hum Gene Ther. 2010 Jul;21(7):903-10. doi: 10.1089/hum.2009.157. PMID 20163245
- [Background] Mah C, Pacak CA, Cresawn KO, Deruisseau LR, Germain S, Lewis MA, Cloutier DA, Fuller DD, Byrne BJ. Physiological correction of Pompe disease by systemic delivery of adeno-associated virus serotype 1 vectors. Mol Ther. 2007 Mar;15(3):501-7. doi: 10.1038/sj.mt.6300100. Epub 2007 Jan 23. PMID 17245350
- [Background] Pacak CA, Conlon T, Mah CS, Byrne BJ. Relative persistence of AAV serotype 1 vector genomes in dystrophic muscle. Genet Vaccines Ther. 2008 Oct 15;6:14. doi: 10.1186/1479-0556-6-14. PMID 18854054
- [Background] Spencer CT, Bryant RM, Day J, Gonzalez IL, Colan SD, Thompson WR, Berthy J, Redfearn SP, Byrne BJ. Cardiac and clinical phenotype in Barth syndrome. Pediatrics. 2006 Aug;118(2):e337-46. doi: 10.1542/peds.2005-2667. Epub 2006 Jul 17. PMID 16847078
- [Background] Smith BK, Collins SW, Conlon TJ, Mah CS, Lawson LA, Martin AD, Fuller DD, Cleaver BD, Clement N, Phillips D, Islam S, Dobjia N, Byrne BJ. Phase I/II trial of adeno-associated virus-mediated alpha-glucosidase gene therapy to the diaphragm for chronic respiratory failure in Pompe disease: initial safety and ventilatory outcomes. Hum Gene Ther. 2013 Jun;24(6):630-40. doi: 10.1089/hum.2012.250. PMID 23570273
- [Background] Smith BK, Martin AD, Lawson LA, Vernot V, Marcus J, Islam S, Shafi N, Corti M, Collins SW, Byrne BJ. Inspiratory muscle conditioning exercise and diaphragm gene therapy in Pompe disease: Clinical evidence of respiratory plasticity. Exp Neurol. 2017 Jan;287(Pt 2):216-224. doi: 10.1016/j.expneurol.2016.07.013. Epub 2016 Jul 21. PMID 27453480
- [Background] Corti M, Elder M, Falk D, Lawson L, Smith B, Nayak S, Conlon T, Clement N, Erger K, Lavassani E, Green M, Doerfler P, Herzog R, Byrne B. B-Cell Depletion is Protective Against Anti-AAV Capsid Immune Response: A Human Subject Case Study. Mol Ther Methods Clin Dev. 2014;1:14033-. doi: 10.1038/mtm.2014.33. PMID 25541616
- [Background] Nathwani AC, Tuddenham EG, Rangarajan S, Rosales C, McIntosh J, Linch DC, Chowdary P, Riddell A, Pie AJ, Harrington C, O'Beirne J, Smith K, Pasi J, Glader B, Rustagi P, Ng CY, Kay MA, Zhou J, Spence Y, Morton CL, Allay J, Coleman J, Sleep S, Cunningham JM, Srivastava D, Basner-Tschakarjan E, Mingozzi F, High KA, Gray JT, Reiss UM, Nienhuis AW, Davidoff AM. Adenovirus-associated virus vector-mediated gene transfer in hemophilia B. N Engl J Med. 2011 Dec 22;365(25):2357-65. doi: 10.1056/NEJMoa1108046. Epub 2011 Dec 10. PMID 22149959
- [Background] Corti M, Cleaver B, Clement N, Conlon TJ, Faris KJ, Wang G, Benson J, Tarantal AF, Fuller D, Herzog RW, Byrne BJ. Evaluation of Readministration of a Recombinant Adeno-Associated Virus Vector Expressing Acid Alpha-Glucosidase in Pompe Disease: Preclinical to Clinical Planning. Hum Gene Ther Clin Dev. 2015 Sep;26(3):185-93. doi: 10.1089/humc.2015.068. PMID 26390092
- [Background] Escolar DM, Henricson EK, Mayhew J, Florence J, Leshner R, Patel KM, Clemens PR. Clinical evaluator reliability for quantitative and manual muscle testing measures of strength in children. Muscle Nerve. 2001 Jun;24(6):787-93. doi: 10.1002/mus.1070. PMID 11360262
- [Background] Barker S, Craik R, Freedman W, Herrmann N, Hillstrom H. Accuracy, reliability, and validity of a spatiotemporal gait analysis system. Med Eng Phys. 2006 Jun;28(5):460-7. doi: 10.1016/j.medengphy.2005.07.017. Epub 2005 Aug 24. PMID 16122966
- [Background] Barker SP, Freedman W, Hillstrom H. A novel method of producing a repetitive dynamic signal to examine reliability and validity of gait analysis systems. Gait Posture. 2006 Dec;24(4):448-52. doi: 10.1016/j.gaitpost.2005.09.008. Epub 2006 Jan 18. PMID 16413189
- [Background] Wary C, Laforet P, Eymard B, Fardeau M, Leroy-Willig A, Bassez G, Leroy JP, Caillaud C, Poenaru L, Carlier PG. Evaluation of muscle glycogen content by 13C NMR spectroscopy in adult-onset acid maltase deficiency. Neuromuscul Disord. 2003 Sep;13(7-8):545-53. doi: 10.1016/s0960-8966(03)00069-5. PMID 12921791
- [Background] Marden FA, Connolly AM, Siegel MJ, Rubin DA. Compositional analysis of muscle in boys with Duchenne muscular dystrophy using MR imaging. Skeletal Radiol. 2005 Mar;34(3):140-8. doi: 10.1007/s00256-004-0825-3. Epub 2004 Oct 22. PMID 15538561
- [Background] Harris RC, Hultman E, Nordesjo LO. Glycogen, glycolytic intermediates and high-energy phosphates determined in biopsy samples of musculus quadriceps femoris of man at rest. Methods and variance of values. Scand J Clin Lab Invest. 1974 Apr;33(2):109-20. No abstract available. PMID 4852173
- [Background] Clark BC, Cook SB, Ploutz-Snyder LL. Reliability of techniques to assess human neuromuscular function in vivo. J Electromyogr Kinesiol. 2007 Feb;17(1):90-101. doi: 10.1016/j.jelekin.2005.11.008. Epub 2006 Jan 19. PMID 16427317
- [Background] Stalberg E, Trontelj JV. The study of normal and abnormal neuromuscular transmission with single fibre electromyography. J Neurosci Methods. 1997 Jun 27;74(2):145-54. doi: 10.1016/s0165-0270(97)02245-0. PMID 9219884